CLINICAL TRIAL: NCT03115528
Title: What is the Difference in the Estimation of Prognosis of Advanced Cancer Patients Between Medical Oncologist, Gynecological Oncologists, and Palliative Care Physicians?
Brief Title: Difference in the Estimation of Prognosis
Status: Withdrawn | Type: Observational
Why Stopped: Terminated at Continuing Review
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-0879
Record Dates: First submitted 2017-04-06; First posted 2017-04-14 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Malignant Neoplasms of Independent (Primary) Multiple Sites
Keywords: Malignant neoplasms of independent (primary) multiple sites; Medical oncologists; Palliative care physicians; Questionnaire; Survey
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical Oncology Physicians: Medical oncology physicians are sent the Estimation of Prognosis questionnaire by email.
  Interventions: Behavioral: Estimation of Prognosis Questionnaire
- Palliative Care Physicians: Palliative care physicians are sent the Estimation of Prognosis questionnaire by email.
  Interventions: Behavioral: Estimation of Prognosis Questionnaire

INTERVENTIONS:
Behavioral: Estimation of Prognosis Questionnaire — Survey will examine two aspects of prognosis estimation: 1.) physician factors, 2.) prognosis estimation and contributing factors to patient prognosis. Survey will take approximately 5 minutes to complete.
  Other Names: Survey

SUMMARY:
Objectives:

Primary Objective:

The primary objective is to identify the difference in the estimation of prognosis of advanced cancer patients between medical oncologists, gynecological oncologists, and palliative care physicians

DETAILED DESCRIPTION:
The goal of this research study is to identify the difference in the estimation of prognosis of advanced cancer patients between medical or gynecological oncologists, and palliative care physicians. Up to 140 patients will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Medical oncologists or gynecological who referred patients to the palliative care team; Palliative Care physicians to whom the patients were referred; Patients with locally advanced, metastatic, or, not curable cancer.
2. 18 years old or older

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical oncologists and palliative care physicians from UT MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Estimation of Patient Overall Survival by Oncologists and by Palliative Care Physicians per Estimation of Prognosis Questionnaire | 6 weeks
  The answer to the question #4, "How long do you think this patient will live?" in the questionnaire is the primary endpoint.
  Denoting the oncologist estimated OS time from the day of palliative care consult to death by TOnc, palliative care physician estimate by TPalliative, and the true OS time by T0, we define the accuracy of the estimation of OS by oncologists and by palliative care physician as ΔOnc = TOnc - T0 ΔPalliative = TPalliative - T0. And the difference between these two estimates is calculated as ΔOS = ΔOnc - ΔPalliative.
  Based on the above formulas, ΔOS is actually calculated as (TOnc- TPalliative). The true survival time, T0, is cancelled out by the subtraction.

CONTACTS AND LOCATIONS:
Overall Officials: Angelique N. Wong, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org